CLINICAL TRIAL: NCT00454194
Title: Phase II Randomized Study of Pemetrexed With Sorafenib Versus Pemetrexed Alone as Second-Line Therapy in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium With or Without Sorafenib as Second-Line Therapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0626; NCI-2009-00657 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000536546 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenosquamous cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Pemetrexed; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral sorafenib tosylate twice daily on days 1-21 and pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pemetrexed disodium; Drug: sorafenib tosylate
- Arm II (Active Comparator): Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pemetrexed disodium

INTERVENTIONS:
Drug: pemetrexed disodium — given IV
Drug: sorafenib tosylate — given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Pemetrexed disodium and sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving pemetrexed disodium together with sorafenib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying pemetrexed disodium and sorafenib to see how well they work compared with pemetrexed disodium alone as second-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with stage IIIB or IV non-small cell lung cancer treated with pemetrexed disodium with or without sorafenib tosylate as second-line therapy.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the tumor response rate and duration of response in patients treated with these regimens.
* Compare the toxicity profile of these regimens in these patients.

Tertiary

* Assess polymorphisms and gene expression in circulating peripheral mononuclear cells and circulating tumor cells of pemetrexed disodium target genes and genes encoding enzymes involved in the transport, activation, and inactivation of pemetrexed disodium.
* Correlate haplotype-tagged single nucleotide polymorphisms or gene expression levels with intracellular levels of pemetrexed disodium polyglutamates, toxicity, and/or efficacy of pemetrexed disodium.
* Assess the expression and polymorphisms in the target genes (i.e., TS, DHFR, GARFT) and methylthioadenosine phosphorylase (as antibodies become available) in paraffin-embedded tissue and compare results to those obtained in circulating tumor tissue, correlating results with response.
* Correlate predictive markers of hypertension (e.g. pharmacogenetics, vascular endothelial growth factor [VEGF]-A, sVEGF receptor-1, and ADMA) with clinical toxicity and outcomes.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1) and North Central Cancer Treatment Group membership. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate twice daily on days 1-21 and pemetrexed disodium IV over 10 minutes on day 1.
* Arm II: Patients receive pemetrexed disodium IV over 10 minutes on day 1. In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected for pharmacokinetic analysis and research studies. Gene expression assays and polymorphism studies (e.g., using polymerase chain reaction) of circulating peripheral blood mononuclear cells are conducted for reduced folate carrier, multidrug resistance-associated protein, folate receptor, BCRP, folylpolyglutamate synthase, MTHFR, methionine synthase, methylthioadenosine phosphorylase, TS, dihydrofolate reductase, GARFT, endothelial nitric oxide synthase, angiotensinogen, dimethylarginine dimethylaminohydrolase, vascular endothelial growth factor (VEGF), and VEGF receptor. Enzyme-linked immunosorbent assays and immunohistochemistry are also conducted.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-squamous cell non-small cell lung cancer (NSCLC)

  * Stage IIIB or IV disease
  * Squamous cell carcinomas are not allowed

    * Adenosquamous histology allowed
* Measurable disease, defined as ≥ 1 lesion with longest diameter ≥ 2.0 cm by conventional techniques or ≥ 1.0 cm by spiral CT scan

  * No nonmeasurable disease only, including small lesions and truly nonmeasurable lesions, including any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* Previously treated with 1 chemotherapy regimen, including adjuvant treatment

  * Prior treatment with adjuvant chemotherapy is allowed and not counted as a regimen
* Symptomatic pleural effusions should be drained prior to study entry

  * No symptomatic serosal effusion (≥ CTCAE v3.0 grade 2 dyspnea) that is not amenable to drainage prior to study entry
* Stable brain metastasis allowed provided the following criteria are met:

  * Treated with either whole brain radiotherapy or gamma knife surgery
  * More than 4 weeks since prior steroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin normal
* Creatinine clearance ≥ 45 mL/min
* AST and ALT ≤ 3 times ULN (5 times ULN if liver has tumor involvement)
* INR < 1.5 OR PT/PTT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after completion of study treatment
* Able to take folic acid, cyanocobalamin, and dexamethasone
* No clinically significant infection
* No known HIV positivity
* No evidence or history of bleeding diathesis or coagulopathy
* No serious nonhealing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No bleeding ≥ grade 2 (except grade 2 petechiae) within the past 4 weeks
* No second primary malignancy except carcinoma in situ of the cervix or nonmelanomatous skin cancer, unless malignancy was diagnosed and definitively treated ≥ 5 years ago with no subsequent evidence of recurrence

  * History of low-grade (Gleason score ≤ 6) localized prostate cancer allowed
  * Patients with a history of DCIS that has been definitively treated will be eligible even if diagnosed < 5 years prior to registration
* No other severe underlying disease or condition that, in the opinion of the investigator, would preclude study compliance or increase risk for serious adverse events
* Able to swallow pills
* No concurrent severe and/or uncontrolled medical conditions, including any of the following:

  * Uncontrolled blood pressure, defined as systolic blood pressure (BP) > 150 mm Hg and/or diastolic BP > 100 mm Hg, in spite of adequate antihypertensive therapy
  * Angina pectoris
  * Congestive heart failure within the past 3 months, unless LVEF > 40%
  * Myocardial infarction within the past 6 months
  * Cardiac arrhythmia
  * Diabetes mellitus
  * Active hemoptysis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy, except for alopecia
* No prior sorafenib tosylate or pemetrexed disodium
* No prior therapy with agents that target VEGF, VEGF receptor, or VEGF receptor tyrosine kinase inhibitor (prior bevacizumab is allowed)
* Prior radiotherapy allowed if all the following criteria are met:

  * No more than 25% of bone marrow was irradiated
  * Measurable disease, whether there is in-field disease progression/recurrence or disease outside the treatment fields of radiation port, is present
* No acetylsalicylic acid dose of ≥ 1.3 grams/day for ≥ 10 days before and after completion of study treatment
* At least 4 weeks since prior full-field radiotherapy
* At least 2 weeks since prior limited-field radiotherapy
* At least 4 weeks since prior major surgery (i.e., laparotomy) or open biopsy
* At least 2 weeks since prior minor surgery
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin C and nitrosoureas)
* At least 2 weeks since prior immunotherapy, biologic therapy, or gene therapy
* At least 4 weeks prior hormonal therapy
* At least 4 weeks since other prior investigational agents
* No concurrent antiretroviral therapy
* No concurrent major surgery
* No concurrent steroids
* No concurrent therapeutic anticoagulation

  * Concurrent prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices allowed provided requirements for PT, INR, or PTT are met
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent grapefruit or grapefruit juice
* No concurrent prophylactic use of colony-stimulating factors
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (207):
- United States (207):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and ten (110) participants were enrolled between October 2007 and April 2010.
Pre-assignment Details: Twelve participants were excluded from all analyses due to five participants had squamous-cell histology, 1 never received treatment and 1 withdrew consent in pemetrexed+sorafenib group; and three participants had squamous-cell histology and 2 never received treatment in pemetrexed alone group.
Groups:
- Arm I (Pemetrexed + Sorafenib): Patients receive oral sorafenib tosylate twice daily on days 1-21 and pemetrexed disodium IV over 10 minutes on day 1.
- Arm II (Pemetrexed): Patients receive pemetrexed disodium IV over 10 minutes on day 1.
Period: Overall Study
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Started | 47 | 51
Completed | 25 | 37
Not Completed | 22 | 14
Not completed — Adverse Event | 7 | 2
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Other Medical Problems | 1 | 2
Not completed — Other Unspecified Reason | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who met the eligibility criteria and started the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed) | Total
Number analyzed (Participants) | 47 | 51 | 98
Age, Continuous [Median (Full Range); unit: years] | 62 [43 to 79] | 62 [49 to 83] | 62 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 27 | 23 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 51 | 98
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 22 | 24 | 46
  1=Symptomatic and fully ambulatory | 25 | 27 | 52
Stage [Count of Participants; unit: Participants] — Stage IIIB: The cancer is continuing to spread from the lungs to the lymph nodes or to nearby structures and organs, such as the heart, trachea and esophagus.> Stage IV: The cancer has metastasized throughout the body and may now affect the liver, bones or brain.
  Participants
    IIIB | 8 | 6 | 14
    IV | 39 | 45 | 84
Prior Bevacizumab [Count of Participants; unit: Participants]
  Yes | 20 | 30 | 50
  No | 27 | 21 | 48
Histology [Count of Participants; unit: Participants]
  Bronchioloalveolar Carcinoma | 1 | 1 | 2
  Adenocarcinoma | 34 | 36 | 70
  Non-small cell lung cancer,not otherwise specified | 10 | 11 | 21
  Large Cell | 2 | 2 | 4
  Large Cell Neuroendocrine | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The progression-free survival (PFS) was defined as the time from date of randomization to the documentation of disease progression or death as a result of any cause, whichever comes first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from randomization to the disease progression or death (up to 5 years)
Population: All participants who met the eligibility criteria and started the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 47 | 51
months | 3.4 [2.6 to 5.7] | 4.1 [1.6 to 5.7]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from study enrollment (randomization) to the time of death from any cause or last follow-up.
Time Frame: Time from randomization to death or last follow-up (up to 5 years)
Population: All participants who met the eligibility criteria and started the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 47 | 51
months | 9.3 [5.9 to 12.2] | 10.4 [7.2 to 13.5]

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from date of randomization to the date at which the patient was removed from the treatment due to progression, toxicity, refusal or other medical problems.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria and ended the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 47 | 50
months | 2.0 [1.5 to 3.1] | 3.1 [1.6 to 5.3]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date at which the patient's earliest best objective status was first noted to be either a complete response (CR) or partial response (PR) to the earliest date progression was documented.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria, have started the study treatment and had confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 6 | 5
months | 7.4 [4.1 to 21.4] | 8.5 [4.7 to 14.4]

5. Secondary Outcome: Number of Participants With at Least One Grade 3 or Above Adverse Events Assessed by NCI CTCAE v4.0
Description: Adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death. The maximum grade for each type of adverse events were recorded for each patient.
Time Frame: Up to 3 years
Population: All participants who met the eligibility criteria and started the treatment.
Measure: Number; unit: participants
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 47 | 51
participants | 43 | 27

6. Secondary Outcome: Confirmed Response Rate (Complete Response and Partial Response) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: A confirmed tumor response was defined as a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 6 weeks apart.
  Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria and started the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Number analyzed (Participants) | 47 | 51
percentage of participants
  Confirmed Response (Partial Response) | 12.8 | 9.8
  Stable Disease | 38.3 | 45.1
  Progression | 23.4 | 35.3
  Not Assessed | 25.5 | 9.8

ADVERSE EVENTS:
Time Frame: Up to 2.6 years
Arm/Group | Arm I (Pemetrexed + Sorafenib) | Arm II (Pemetrexed)
Serious Adverse Events (participants affected / at risk) | 13/47 | 7/51
Other Adverse Events (participants affected / at risk) | 47/47 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pemetrexed + Sorafenib) (N=47) | Arm II (Pemetrexed) (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 2 (2)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pemetrexed + Sorafenib) (N=47) | Arm II (Pemetrexed) (N=51)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 42 (208) | 42 (218)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (6) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (5)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (5)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (6) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (2)
Watering eyes (Eye disorders) | 3 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 19 (33) | 15 (28)
Constipation (Gastrointestinal disorders) | 7 (10) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 23 (68) | 14 (19)
Dry mouth (Gastrointestinal disorders) | 2 (13) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 14 (27) | 3 (5)
Flatulence (Gastrointestinal disorders) | 2 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 20 (42) | 8 (12)
Nausea (Gastrointestinal disorders) | 31 (87) | 24 (83)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (44) | 12 (28)
Chest pain (General disorders) | 3 (4) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (2) | 2 (7)
Fatigue (General disorders) | 46 (246) | 48 (228)
Fever (General disorders) | 9 (12) | 6 (8)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 2 (4) | 2 (2)
Pain (General disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (5)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 2 (3) | 1 (3)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (22) | 3 (4)
Alkaline phosphatase increased (Investigations) | 7 (18) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 6 (48) | 1 (1)
Cardiac troponin I increased (Investigations) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (3)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 29 (87) | 18 (41)
Lipase increased (Investigations) | 4 (9) | 6 (8)
Lymphocyte count decreased (Investigations) | 8 (39) | 3 (19)
Neutrophil count decreased (Investigations) | 21 (40) | 12 (23)
Platelet count decreased (Investigations) | 20 (52) | 14 (20)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 21 (46) | 14 (50)
Anorexia (Metabolism and nutrition disorders) | 28 (70) | 25 (61)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (21) | 8 (45)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (5) | 4 (12)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (5) | 1 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 17 (37) | 11 (33)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (19) | 5 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 1 (3)
Dizziness (Nervous system disorders) | 2 (2) | 1 (2)
Headache (Nervous system disorders) | 5 (5) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (96) | 23 (117)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 6 (9) | 1 (11)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (24) | 7 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (24) | 11 (21)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (19) | 1 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 23 (72) | 1 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 14 (19) | 4 (6)
Rash desquamating (Skin and subcutaneous tissue disorders) | 21 (33) | 4 (6)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 19 (56) | 11 (29)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less